CLINICAL TRIAL: NCT06289049
Title: Feasibility and Preliminary Efficacy of Heavy Lifting Strength Training Versus Usual Care in Head and Neck Cancer Survivors: A Randomized Controlled Trial
Brief Title: Heavy Strength Training in Head and Neck Cancer Survivors
Acronym: LIFTING2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HREBA.CC-24-0021
Record Dates: First submitted 2024-02-22; First posted 2024-03-01 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Head and Neck Neoplasms; Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma; Head and Neck Carcinoma
Keywords: Strength Training; Exercise; Quality of Life; Randomized Controlled Trial
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Motor Activity

STUDY DESIGN:
Masking Description: Participants and investigators will not be blinded to group assignment given the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): The exercise intervention will consist of 24 supervised, heavy lifting strength training exercise sessions over a 12 week period. The exercise frequency will be two times per week. Main exercises will consist of barbell back squat, bench press, and dead lift.
  Interventions: Other: Experimental
- Usual Care Group (No Intervention): Participants randomized to the usual care group will be asked to continue will their typical daily routine during the 12 week study period, and not begin any new exercise program to increase their exercise levels from baseline. They will not receive any information or education regarding exercise. After the postintervention assessments, participants in the usual care group will be offered a 4-week introduction to heavy lifting strength training program and/or referred to a community-based exercise program

INTERVENTIONS:
Other: Experimental — Three primary exercises will be included in the exercise sessions for participants randomized to this group: barbell back squat, bench press, and dead lift
  The weight will be progressively increased overtime based on participants' perceived exertion and repetitions in reserve. Number of repetitions performed for each exercise will begin at 10 repetitions in weeks 1-2, with gradual progression to lifting heavier loads of 3-5 sets of 1-5 repetitions between weeks 6-12.
  Other Names: Exercise Group
  Arms: Exercise Group

SUMMARY:
Despite improvements in treatments, head and neck cancer survivors (HNCS) still endure acute and chronic side effects such as loss of muscular strength, limitations in physical functioning, fatigue, and swallowing difficulties that impact quality of life (QoL) and limit return to work. Light-to-moderate intensity strength training (LMST) has been shown to improve some side effects. Heavy lifting strength training (HLST) may further improve outcomes in some populations, however, only one small pilot study has focused on HNCS. The LIFTING 2 trial will be the first to examine the feasibility and effects of a HLST program versus no exercise in HNCS.

DETAILED DESCRIPTION:
1. Background and Rationale

   Despite improvements in treatments, head and neck cancer survivors (HNCS) still endure acute and chronic side effects such as loss of muscular strength, limitations in physical functioning, fatigue, and swallowing difficulties that impact quality of life (QoL) and limit return to work. Light-to-moderate intensity strength training (LMST) has been shown to improve some side effects. Heavy lifting strength training (HLST) may further improve outcomes in some populations, however, only one small pilot study has focused on HNCS.
2. Research Question & Objectives

   The primary aim of the proposed study is to further establish the feasibility of HLST in HNCS which will be based on the eligibility rate, recruitment rate, one-repetition max (3RM) testing rate, HLST program adherence, and follow-up assessment rate. A secondary aim is to provide preliminary evidence of the effects of a HLST program compared to usual care (UC) in HNCS. The primary efficacy outcome will be upper and lower muscular strength assessed by reliable 3-repetition maximum (3RM) tests on the chest press and leg press machines. Secondary efficacy outcomes include physical function, handgrip strength, body composition, QoL, fear of cancer recurrence, symptom burden, pain, anxiety, fatigue, stress, self-esteem, shoulder mobility, sleep, malnutrition status, and swallowing abilities.
3. Methods

This single-centre, two-armed, randomized controlled trial will recruit 60 HNCS ≥1-year posttreatment, and randomly assign them to the HLST group or UC group. For the HLST group, the 12-week exercise intervention will include supervised training 2 days per week. The HLST group will progress to lifting low repetitions of heavy loads at 80-90% of one repetition maximum (1RM), whereas the UC group will not receive any exercise prescription or instruction during the 12-week intervention, but will be offered a 4-week introduction to HLST program and/or referred to a community-based program after the postintervention assessments are complete. Assessments for both groups will occur at baseline and postintervention and include reliable 3RM strength tests, bioelectrical impedance analysis (BIA), Senior's Fitness Test, and validated QoL questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* males and females, 18 years of age and older
* any head and neck cancer subtype, stage, and treatment type
* at least 1-year posttreatment with adequate shoulder range of motion (must meet minimum cutpoints for active flexion and abduction to be eligible)
* no unmanaged medical conditions, alcohol, or drug abuse
* approved for exercise by oncologist and a certified exercise physiologist or kinesiologist
* ability to understand and communicate in English

Exclusion Criteria:

* has met the Canadian Physical Activity strength training guidelines within the past one-month: at least two days per week of muscle and bone strength training activities using major muscle groups
* currently involved in a different exercise trial or clinical drug trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Baseline, postintervention (12 weeks), and monitored throughout 12 week study period
  Recruitment range: 40 to 60 participants; Higher=better and more available data
Adherence to a heavy lifting strength training program | Baseline, postintervention (12 weeks), and monitored throughout 12 week study period
  Adherence rate: 0 to 100 percent of exercise sessions; Higher=better
Completion of maximal strength testing | Baseline and postintervention (12 weeks)
  3 repetition maximum testing rate: 0 to 100 percent; Higher=better
Followup assessment rate | Postintervention (12 weeks)
  Followup assessment rate: 0 to 100 percent; Higher=better
Safety | Baseline, postintervention (12 weeks), and monitored throughout 12 week study period
  Adverse events: minimum: no adverse events, maximum: no maximum. Higher=worse

SECONDARY OUTCOMES:
Muscular Strength | Baseline and Postintervention (12 weeks)
  Assessed via 3 repetition maximum tests on the chest press and leg press machines
  Minimum: 0 kilograms, Maximum: none. Higher score=better strength
Cancer Specific Quality of Life | Baseline and Postintervention (12 weeks)
  Assessed via cancer specific European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire
  Minimum: 0 points, Maximum: 100 points. Higher score=better quality of life
Fear of Cancer Recurrence | Baseline and Postintervention (12 weeks)
  Assessed via the Fear of Cancer Recurrence Inventory - Short Form
  Minimum: 0 points, Maximum: 36 points. Higher score=worse fear of cancer recurrence
Symptom Burden | Baseline and Postintervention (12 weeks)
  Assessed via the revised Edmonton Symptom Assessment System
  Minimum: 0 points, Maximum: 100 points. Higher score=worse cancer symptoms
Perceived Stress | Baseline and Postintervention (12 weeks)
  Assessed via the Perceived Stress Scale
  Minimum: 0 points, Maximum: 56 points. Higher score=worse perceived stress
Self-Esteem | Baseline and Postintervention (12 weeks)
  Assessed via the Rosenberg Self-Esteem Scale
  Minimum: 10 points, Maximum: 40 points. Higher score=better self-esteem
Sleep Habits | Baseline and Postintervention (12 weeks)
  Assessed via the Insomnia Severity Index
  Minimum: 0 points, Maximum: 28 points. Higher score=worse insomnia
Malnutrition Status | Baseline and Postintervention (12 weeks)
  Assessed via the Patient Generated Subjective Global Assessment with reference to the Global Leadership Initiative on Malnutrition
  Minimum: 0 points, Maximum: 36 points. Higher score=worse, high risk of malnutrition
  0-1 points: no intervention required at this time. Re-assessment on routine and regular basis during treatment.
  2-3 points: patient & family education by dietitian, nurse, or other clinician with pharmacologic intervention as indicated by symptom survey and lab values as appropriate
  4-8 points: requires intervention by dietitian, in conjunction with nurse or physician as indicated by symptoms
  ≥ 9 points: indicates a critical need for improved symptom management and/or nutrient intervention options
Swallowing Abilities | Baseline and Postintervention (12 weeks)
  Assessed via the MD Anderson Dysphagia Inventory
  Minimum: 20 points, Maximum: 100 points. Higher score=better swallowing ability
Shoulder Range of Motion | Baseline and Postintervention (12 weeks)
  Assessed via seated active flexion and abduction using a goniometer
  Minimum: 150 degrees (18-50 years); 130 degrees (over 50 years), Maximum: none Higher score=better shoulder mobility
Body composition | Baseline and Postintervention (12 weeks)
  Assessed via bioelectrical impedance analysis (InBody 770)
  Minimum: none, Maximum: none. Higher score=variable Higher fat free mass score=better Higher fat mass score=worse
Handgrip Strength | Baseline and Postintervention (12 weeks)
  Assessed via held held dynamometer
  Minimum: 0 kilograms, Maximum: none. Higher score=better hand grip strength
Physical Function | Baseline and Postintervention (12 weeks)
  Assessed via the six minute walk test
  Minimum: 0 metres, Maximum: none. Higher score=better physical function

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Courneya, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No